CLINICAL TRIAL: NCT04324983
Title: Identification of Predictive Biomarkers for Successful Salvage Surgeries on PSMA-PET-positive Limited Metastatic Prostate Cancer Relapses
Brief Title: Identification of Predictive Biomarkers
Acronym: BioPoP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martini-Klinik am UKE GmbH (Other)
Collaborators: Erich und Gertrud Roggenbuck-Stiftung zur Förderung der Krebsforschung (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BioPoP-MK-2020-2
Record Dates: First submitted 2020-03-03; First posted 2020-03-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer Recurrent
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: In this single-arm prospective clinical study, various blood- and serum-based biomarkers, from patients with early PSMA PET positive limited metastatic prostate cancer relapse after radical prostatectomy, will be examined according to their potential predictive significance for a successful salvage surgery. Results from the various biomarker values, after salvage surgery, with following clinical endpoints will be assessed:
  1. postoperative complete biochemical response (cBR: PSA <0,2ng/ml)
  2. biochemical relapse-free without further prostate cancer specific treatment (time from salvage surgery to first PSA level >0,2ng/ml)
  3. prostate cancer specific treatment-free interval (time from salvage surgery to initiation of a prostate cancer specific treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomarker (Other): This single-arm study is a Phase I study to exploratively identify potential biomarkers in patients with early prostate cancer relapse and limited metastases in PSMA-PET, who need further assistance in treatment decisions (for or against local treatment options).
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Additional blood sample of about 30 ml that will be drawn for biomarker analyses (2 EDTA = ethylenediaminetetraacetic acid and 1 Cell-search-tubes).The drawn blood for CTC-Analysis and biomarker identification will be promptly processed ac-cording to the established standards at the Institute for Tumor Biology (see below).
  The histological analysis of the resected tissue during salvage surgery is carried out according to clinical routine (conventional haematoxylin and eosin stained and PSMA-Immunohistochemistry). Additionally, tissue samples will undergo molecularpathological analysis if this does not affect routine pathological examination.

SUMMARY:
Molecular nuclear imaging in prostate cancer has made significant progress in the last few years. The introduction of tracers that target the prostate-specific membrane antigen (PSMA) has profoundly influenced imaging diagnostics in prostate cancer. In case of relapse after curative treatment (especially after radical prostatectomy), PSMA positron emission tomography (PET) has the ability to detect lesions already at very low prostate-specific antigen (PSA) levels. The improved detection of relapses increases the interest of individualized targeted therapies in patients with prostate cancer recurrence. Thus, this development led to the acceptance of PSMA PET for diagnostics in prostate cancer patients with biochemical relapses in national and international guidelines.

DETAILED DESCRIPTION:
As mentioned before, current data on salvage lymphadenectomy in prostate cancer is very limited and stems mainly from retrospective series. Prospective studies are not available. Furthermore, most of these analyses are based on choline-based positron emission tomography, which by now has been progressively replaced with the significantly more sensitive and specific PSMA-based PET. Diagnostic advantages are especially obvious in early biochemical recurrence with low PSA levels . The high specificity of a PSMA Tracer in diagnosing prostate cancer tissue is further demonstrated by the introduction of PSMA-radioguided surgery. Here, patients are injected intravenously before surgery with 111In- or 99mTc-labeled PSMA ligands in order to enhance intraoperative detection of affected lymph nodes that show radiotracer accumulation.

Regarding biomarkers used in prostate cancer, besides PSA and PSA-associated variations, there also exists a multiple number of different biomarkers. However, most of these biomarkers are used in the primary diagnostic setting or in advanced metastatic tumor stages with a castration-resistant stage. However, especially in early biochemical recurrences there is a need for biomarkers to help determine whether or not local salvage treatment can or should be considered. Circulating tumor cells (CTCs) are promising candidates as a biomarker, that could support the decision-making process. While the prognostic relevance of CTCs for patients with a metastatic castration-resistant stage prostate cancer has been shown in many studies, far less data exists for patients with hormone-sensitive metastatic prostate cancer. Regardless of the fact, survival is associated with the number of CTCs measured in peripheral blood. Recently, we were able to show that CTCs in patients with limited metastatic prostate cancer exhibited higher prognostic relevance, before and after cytoreductive radical prostatectomy, than conventional biomarkers (PSA, LDH =lactate Dehydrogenase and BAP). Even when the conventional biomarkers were combined with routine markers and CTCs, the prognostic relevance did not increase. Although the case numbers were very small, in the future, CTCs could still help identify patients that would most profit from a cytoreductive radical prostatectomy.

Therefore, this project will investigate whether or not CTCs can preoperatively provide prognostic information on the postoperative oncological response, as described in the study protocol. The plan is to withdraw blood (7,5 ml) before surgery from 150 limited metastatic prostate cancer patients. These patients have to qualify for salvage surgery according to the PSMA-PET. The blood will be examined with the Cell-Search-Systems for CTCs and their PSMA Expression.

Plasma samples and peripheral blood mononuclear cells (PBMCs) from peripheral blood will also be stored. These samples will be used later for a further project on prostate cancer-specific exosomes where PSMA positivity and cell-free circulating nucleic acids will be examined. The expertise for such analyses, standard operating procedures (SOPs) and necessary equipment are available.

Furthermore, the Institute for Tumor Biology has recently established a new blood test for detecting breast cancer. This test will also be used on prostate cancer patients within the scope of this project. This test measures the serum concentration of Cyr61-Proteins. The Institute has established an Enzyme-Linked Immunosorbent Assay (ELISA), which has already been successfully implemented for the analysis of blood plasma in 527 breast cancer patients. Consequently, this newly developed blood test presents an important improvement in the diagnosis of breast cancer (International patent System 2018/054052). It would also like to test this method for its adequacy and improvement in the diagnosis of prostate cancer within the context of this project.

Furthermore, in a subset of patients additionally tissue from metastatic lymph nodes will be collected for molecularpathologic analysis if tissue sampling does not affect routine pathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good general health and an expected life expectancy of > 10 years
* Diagnosis of prostate cancer relapse
* Evidence of positive lymph nodes or soft tissue metastases as seen in PSMA PET

Exclusion Criteria:

* Contraindication for a surgical procedure
* Clinical suspicion of systemic disease as determined by PSMA PET
* PSMA PET examination older than 4 months at time of surgery

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Rate of complete biochemical response (cBR: PSA <0,2ng/ml) | 6 months
  PSA Level after salvage lymphadenectomy without adjuvant prostate cancer-specific treatment

SECONDARY OUTCOMES:
Prostate cancer-specific treatment-free survival after salvage surgery | 3, 6, 12 and 24 months
  PSA-Level after salvage lymphadenectomy
Questionnaire Quality of life | 3, 6, 12 and 24 months
  Expanded prostate cancer index Composite (EPIC 26)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Maurer, Prof., Principal Investigator — Head Doctor
Locations (1):
- Martini-Klinik am UKE GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No